CLINICAL TRIAL: NCT03282266
Title: A Randomised, Single-blind, Sham Operation-controlled Study to Evaluate the Safety and Efficacy of the Pulmonary Artery Denervation for the Treatment of Pulmonary Arterial Hypertension
Brief Title: Safety and Efficacy of Pulmonary Artery Denervation in Patients With Pulmonary Arterial Hypertension
Acronym: PADN-CFDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Pulnovo Medical (Wuxi) Co., Ltd. (Industry); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tianjin Medical University General Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Beijing Anzhen Hospital (Other); Shenyang Northern Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Hang Zhang, Vice Director of Cardiovascular Department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20170501
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant
Masking Description: sham operation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PADN + 5-phosphodiesterase (Experimental): A total of 64 patients are assigned to PADN + 5-phosphodiesterase group after randomization schedule.
  Interventions: Procedure: PADN
- Sham operation + 5-phosphodiesterase (Sham Comparator): A total of 64 patients are assigned to sham operation + 5-phosphodiesterase group after randomization schedule.
  Interventions: Procedure: Sham operation

INTERVENTIONS:
Procedure: PADN — PADN was performed at three sites at the conjunctional area between the distal main trunk and the ostial left branch. The following ablation parameters were programmed at each point: a temperature of 45 ℃-50 ℃, energy ≤15 W, and a time of 120 seconds. The procedure would cease for 10 seconds if the patient felt intolerable chest pain during the procedure. The EKG and pressure lines (including cardiac output) were monitored and continuously recorded throughout the procedure.
  Other Names: pulmonary artery denervation
  Arms: PADN + 5-phosphodiesterase
Procedure: Sham operation — The radiofrequency ablation catheter placed, no ablations for patients in the sham PADN group.
  Arms: Sham operation + 5-phosphodiesterase

SUMMARY:
The objective of this randomized control trial is to gain clinical insight on the use of pulmonary artery denervation (PADN) for the treatment of pulmonary arterial hypertension (PAH). The primary objective is to assess effectiveness and safety of PADN for the treatment of PAH.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the change in 6-minute walk distance (6MWD) of PADN on PAH patients. Based on the previous studies, the 6MWD was 13±24 m after 6-month treatment using target drugs. And our previous data showed that 6MWD at 6-month after PADN procedure was 65±85 m. As a result, a total of 128 patients with Group I PAH are randomized at a ratio of 1:1 to either PADN procedure plus phosphodiesterase-5 inhibitors (PDE5i) group (PADN group) or sham-PADN procedure plus PDE5i group (Sham group) using a randomization schedule blocked by site. The combination therapy of PDE5i with additional other PAH-specific target drugs is not recommended for all patients and is left at physician's discretion in both groups.

ELIGIBILITY:
Inclusion Criteria:

Provision of informed consent prior to any study specific procedures; Men and women 18 years and older; Group I PAH, defined as a mPAP≥25mmHg, PCWP<15mmHg and PVR[The PVR =(mPAP-PCWP)/CO]>3.0 Woods unit.

Exclusion Criteria:

General exclusion criteria:

Pregnancy and breast feeding mother; Estimated life expectancy < 12 months; Scheduled major surgery in the next 6 months; Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk; Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 30 days.

Procedural exclusion criteria:

WHO group II, III, IV, V PH Severe Renal dysfunction (Ccr<30 ml/min) Blood platelet count<100,000/L Expected life span<6-month Systematical inflammation Malignant cancer(s) Tricuspid valve stenosis, Supra-pulmonary valve stenosis Allergic to studied drugs or metal materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in 6-Minute Walk Distance (6MWD) at 6 Month | Baseline, 6 Month
  6MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.

SECONDARY OUTCOMES:
Change From Baseline in Systolic Pulmonary Arterial Pressure (sPAP) at 6 Month | Baseline, 6 Month
  sPAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position.
Change From Baseline in Mean Pulmonary Arterial Pressure (mPAP) at 6 Month | Baseline, 6 Month
  mPAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position.
Change From Baseline in Cardiac Output (CO) at 6 Month | Baseline, 6 Month
  CO is the volume of blood being pumped by the heart ventricle in the time interval of one minute.
Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at 6 Month | Baseline, 6 Month
  PCWP was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure.
Change From Baseline in Pulmonary Vascular Resistance (PVR) at 6 Month | Baseline, 6 Month
  PVR: calculated by subtracting PCWP from mPAP and dividing by cardiac output in pulmonary circulation (COpulm).
Change From Baseline in Right Ventricle Functional at 6 Month | Baseline, 6 Month
  Right ventricle functional measures by echocardiography include right ventricle systolic and diastolic functional variables.
PAH-related events | 6 Month
  PAH-related events were defined as those caused by worsening of PAH, initiation of treatment with intravenous or subcutaneous prostanoids, lung transplantation, atrial septostomy, or all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Hang Zhang, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SL, Zhang FF, Xu J, Xie DJ, Zhou L, Nguyen T, Stone GW. Pulmonary artery denervation to treat pulmonary arterial hypertension: the single-center, prospective, first-in-man PADN-1 study (first-in-man pulmonary artery denervation for treatment of pulmonary artery hypertension). J Am Coll Cardiol. 2013 Sep 17;62(12):1092-1100. doi: 10.1016/j.jacc.2013.05.075. Epub 2013 Jul 10. PMID 23850902
- [Background] Chen SL, Zhang H, Xie DJ, Zhang J, Zhou L, Rothman AM, Stone GW. Hemodynamic, functional, and clinical responses to pulmonary artery denervation in patients with pulmonary arterial hypertension of different causes: phase II results from the Pulmonary Artery Denervation-1 study. Circ Cardiovasc Interv. 2015 Nov;8(11):e002837. doi: 10.1161/CIRCINTERVENTIONS.115.002837. PMID 26553699
- [Derived] Zhang H, Wei Y, Zhang C, Yang Z, Kan J, Gu H, Fan F, Gu H, Wang Q, Xie D, Zhang G, Guo X, Yin Y, Jin B, Zhou H, Yang Z, Wang Z, Xin Y, Zhang C, Meng L, Wang X, Sun J, Zhao C, Zhang J, Yan X, Chen F, Yao C, Stone GW, Chen SL. Pulmonary Artery Denervation for Pulmonary Arterial Hypertension: A Sham-Controlled Randomized PADN-CFDA Trial. JACC Cardiovasc Interv. 2022 Dec 12;15(23):2412-2423. doi: 10.1016/j.jcin.2022.09.013. Epub 2022 Sep 18. PMID 36121246